CLINICAL TRIAL: NCT04411589
Title: Evaluation of the Diagnostic Ability of White Light Endoscopy and Magnifying Endoscopy With Optical Enhancement System in Early Gastric Cancer and Intraepithelial Neoplasia: a Prospective Randomized Controlled Trial
Brief Title: The Diagnostic Ability of White Light Endoscopy and Magnifying Endoscopy With Optical Enhancement System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, doctoral supervisor of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2018SDU-QILU-125
Record Dates: First submitted 2020-05-24; First posted 2020-06-02 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Early Gastric Cancer
Keywords: Early gastric cancer, Optical enhancement system
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnifying endoscopy with optical enhancement system group (Experimental): Patients in this group go through gastroscopy under the magnifying endoscopy with optical enhancement system.
  Interventions: Device: magnifying endoscopy with optical enhancement system
- white light endoscopy group (Active Comparator): Patients in this group go through gastroscopy under white light endoscopy.
  Interventions: Device: white light endoscopy system

INTERVENTIONS:
Device: magnifying endoscopy with optical enhancement system — A complete screening examination was first performed with white light endoscopy. Additionally, the types of endoscopic GIN and EGC were recorded according to the Paris Classification. After visualization in white light mode, the stomach was reinspected by using OE mode2. Then, in vivo diagnoses of lesions were made by using OE mode1 according to VS theory. For all suspicious areas, a minimum of one biopsy specimens were first taken in a targeted fashion.
  Arms: Magnifying endoscopy with optical enhancement system group
Device: white light endoscopy system — A complete screening examination was first performed with white light endoscopy. Additionally, the types of endoscopic GIN and EGC were recorded according to the Paris Classification. For all suspicious areas, a minimum of one biopsy specimens were first taken in a targeted fashion.
  Arms: white light endoscopy group

SUMMARY:
The purpose of this study is to valuation of the diagnostic ability of white light imaging and magnifying endoscopy with optical enhancement system in early gastric cancer and intraepithelial neoplasia.

DETAILED DESCRIPTION:
Stomach cancer is the second most common cause of cancer death. Endoscopic identification and treatment of gastric intestinal metaplasia (GIM) and early gastric cancer (EGC) is essential to improve patients' 5-year survival rates. Conventional endoscopy with white light imaging (WLI) is widely used for endoscopic evaluation of EGCs. However, conventional endoscopic visualization of EGCs has a high rate of interobserver variability and correlates poorly with the histological findings. For this reason, diagnosis has been based mostly on repeated endoscopy with multiple biopsy samples. It has been reported that optical enhancement (OE) system is useful for discriminating cancerous lesions from non-cancerous lesions. The OE system is the newly developed image-enhanced endoscopic technology, which combines high definition white light endoscopy (WLE) and optical filters that limit the spectral characteristics of the illumination light. The optical filters can achieve higher overall transmittance by connecting the peaks of the hemoglobin absorption spectrum creating a continuous wavelength spectrum. Magnifying endoscopy is useful for observing the mucosal structures and microvessels. The VS theory proposed by Yao K is widely used in Magnifying endoscopy with optical enhancement system (ME-OE). Based on technical considerations, it is conceivable that ME-OE imaging techniques might have a distinct advantage over WLE in the diagnosis of endoscopic lesions. However, few reports have objectively proved that ME-OE is superior to WLE in the detection rate and diagnostic efficiency of EGCs.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years with H. pylori infection or histologically verified gastric lesions (chronic atrophic gastritis, intestinal metaplasia, GIN or EGC)
* Or patients aged 40-80 years from a region with high incidence of gastric cancer
* Or patients aged 40-80 years with first-degree relative of patients with gastric cancer
* Or patients aged 40-80 years with high-risk factors for gastric cancer (high salt or pickle diet or smoking or heavy drinking)

Exclusion Criteria:

* A history of gastrectomy
* Active gastrointestinal bleeding or advanced gastric carcinoma
* Coagulopathy or severe underlying diseases
* Pregnancy or lactation
* Absence of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
detection rate of GIN and EGC | 3 months
  The primary outcome was the detection rate of gastric intestinal metaplasia (GIM) and early gastric cancer (EGC) in a per-patient analysis.

SECONDARY OUTCOMES:
sensitivity, specificity of diagnostic performances of GIN and EGC | 3 months
positive predictive value of diagnostic performances of GIN and EGC | 3 months
negative predictive value of diagnostic performances of GIN and EGC | 3 months
diagnostic accuracy in a per-biopsy analysis | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Principal Investigator — Shandong University Qilu hosipital, China
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Derived] Wan M, Li GC, Ma MJ, Liu J, Li Z, Zuo XL, Li YQ. Optical enhancement with magnification versus white-light endoscopy for detecting gastric intestinal metaplasia and neoplasia: a randomized controlled trial. Gastrointest Endosc. 2025 Sep;102(3):337-344.e1. doi: 10.1016/j.gie.2025.02.015. Epub 2025 Feb 15. PMID 39956464